CLINICAL TRIAL: NCT03891147
Title: A Randomized, Single-blind, Controlled Trial of Electroacupuncture for the Treatment of Symptomatic Gallstone Diseases
Brief Title: A Clinical Trial of Electro-acupuncture for Treating Gallstone Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Wendy Wong, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMRF-13141331
Record Dates: First submitted 2019-02-13; First posted 2019-03-26 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Gallstones
Keywords: symptomatic gallstone diseases; electro-acupuncture
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Intervention Model Description: A two arm pragmatic randomized controlled trial design will be conducted at the Prince of Wales Hospitals. 132 patients diagnosed of symptomatic gallstone diseases are on waiting list for cholecystectomy or being recommended to have cholecystectomy by surgeons will be allocated in either EA group (n = 66); or control group (n=66). Treatment group will be offered 20 sessions of EA in 10 weeks, while the control group will remain in the usual care for solely assessment. Primary outcome is the proportion of patients with total clearance of gallstones after treatment with confirmation by ultrasonography. The secondary outcome is the monitoring the incidence of common bile duct stone by liver function test (LFT) and MRCP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electro-acupunture (EA) group (Experimental): Patients will receive the treatment of electro-acupuncture with acupoints (i) Riyue (GB-24) ; (2) Danshu (B19) ; (3) Ganshu (B18) ; (4) Qimen (LR14) ; (5) Yanglingquan (GB34)
  The EA will be conducted by using disposable acupuncture needles (0.30 mm in diameter and 25-40 mm in length). The needles are inserted at a depth of 10-30 mm vertically or obliquely into acupoints, on which electrical stimulation with continuous waves with 2 Hz and 100 Hz are delivered for 15 min for each frequency through an electrical acupuncture treatment instrument (Hwarto, SDZ-II). The intensities of stimulation are adjusted to a level at which patients feel most comfortable. Each session lasts for 30 minutes.
  Interventions: Other: Electro-acupuncture
- Usual care group (No Intervention): Participants randomized to usual care will continue regular follow up arranged by their visiting physicians in public or private sectors. Current usual care of these patients is limited to symptomatic treatment and dietary advice only during the follow-up session in out-patient clinic until the end of observation period (week 10).

INTERVENTIONS:
Other: Electro-acupuncture
  Arms: Electro-acupunture (EA) group

SUMMARY:
Background: Electro-acupuncture (EA) is commonly used as an alternative treatment for gallstone disease. This study aimed to investigate the effectiveness of EA. If shown effective, patients could preserve their gallbladders from cholecystectomy.

Methods: Within a treatment period of 10 weeks, 132 subjects with symptomatic gallstone diseases (size <=8mm) were randomly allocated into either treatment group (n=66), or control group (n=66). Treatment group was offered 20 EA sessions while the control group were clinically observed. The primary outcome was the proportion of patients with total/partial clearance of gallstone confirmed by ultrasonography between the two groups. Secondary outcomes were the evaluation of Patients Reported Outcomes (PROs) (e.g.SF6D, GIQLI) collected throughout the treatment period.

DETAILED DESCRIPTION:
Introduction:

Gallstone disease is a significant health problem affecting 10%-15% of the adult population. Gallstone diseases include cholelithiasis, choledocholithiasis or intrahepatic gallstones. In Hong Kong, gallstones are found in 2-3% of the population and 20% of the gallstones are symptomatic. To date, cholecystectomy is the gold standard treatment for acute cholecystitis. Laparoscopic cholecystectomy is the preferred modality for elective cholecystectomy and is advised mainly for symptomatic gallstones such as acute cholecystitis or biliary pancreatitis. It is recommended that the cholecystectomy should be performed within weeks after resolution of any episode of complications. However, in Hong Kong, the average waiting time for cholecystectomy ranged from 9 months to years. The prolonged waiting time increases the risk of severe complications such as high conversion rate of acute inflammation, pancreatitis, cholecystitis; obstructive jaundice or gallbladder cancer.

Acupuncture has been extensively applied in clinical practice to treat symptomatic gallstone diseases in the ancient Traditional Chinese Medicine (TCM) diagnoses of hypochondrite pain , jaundice or pyretic thoracic retention. The mechanism of acupuncture had been studied with (1) increasing of the excretory function of gall bladder; (2) increasing the relaxation of the sphincter of Oddi and (3) increasing the secretion of bile. All the above actions aim at promoting the spontaneous clearance of gallstones from the biliary system to the gut. In fact, gallstone clinic are commonly available in acupuncture department of Chinese Medicine Hospitals in China for daily practice. Owing to the poor clinical trial methodology, the evidence of effectiveness of acupuncture were not well established yet.

As a highly recognized traditional therapy, acupuncture has been increasingly used for the treatment of pain. Early studies in both animals and human subjects found that electroacupuncture (EA) stimulation on certain acupoints could induce the release of endogenous opioid peptides and modulate the activities of related receptors in the brain. These opioid peptides mainly include endomorphin, β-endorphin, enkephalins, and dynorphin. Furthermore, EA stimulation also could modulate central neurotransmitters, including serotonin and dopamine, which play important roles in pain signal processing. In addition, it was found that EA can help antagonize smooth muscle relaxation. Based on these findings, EA may be useful in fostering the expelling effect of the smooth muscle of the gallbladder.

There had been case reports and case series supporting the use of EA in the treatment of symptomatic gallstones. However, only one controlled trial has reported EA in treating gallstone diseases on 120 patients with total excretion of gallstones with confirmed with ultrasonography (Treatment group 30% vs control group 16.7%, p<0.05) with stone size smaller than 1cm. However, this study did not report any adverse event during the course of treatment. Apart from absence of adverse events reporting, the reference study did use the percentage of patients with total excretion of gallstone confirmed by ultrasound scanning as the primary outcome. Bearing in mind safety as the first priority, the study did not adopt any blinding in the clinical trial and could overestimate the effectiveness of acupuncture in treating gallstone diseases. With our proposed rigorous conduction of clinical trial in terms of objective assessment of primary outcome and the blinding of assessor, the investigators hope to confirm the effectiveness of acupuncture in gallstone diseases despite of the results published in China. In fact, many patients in Hong Kong are waiting for cholecystectomy with average time of 9 months to years owing to the less urgency of the operation. The investigators hope this study could confirm the effectiveness of acupuncture on gallstone diseases so as to develop more evidence. To substantiate the effectiveness and safety of EA as an alternative intervention for symptomatic gallstones in clinical practice, this study aims at pioneering a well-designed, long-term, large-scale controlled trial for further evaluation of the effectiveness of EA in treating gallstone diseases.

Aims: to evaluate the effectiveness and safety of EA as an alternative treatment in symptomatic gallstone diseases. Based on the pragmatic nature of the trial, this study will also explore the health economic evaluation of additional acupuncture services against usual care.

Methods: A two arm pragmatic randomized controlled trial design will be conducted at the Prince of Wales Hospitals. 132 patients diagnosed of symptomatic gallstone diseases are on waiting list for cholecystectomy or being recommended to have cholecystectomy by surgeons will be allocated in either EA group (n = 66); or control group (n=66). Treatment group will be offered 20 sessions of EA in 10 weeks, while the control group will remain in the usual care for solely assessment. Primary outcome is the proportion of patients with total clearance of gallstones after treatment with confirmation by ultrasonography. The secondary outcome is the monitoring the incidence of common bile duct stone by liver function test (LFT) and MRCP.

Implication of this study The most expected and clinically significant findings should be the exploratory effectiveness of EA that promotes the excretion of the gallstones. In addition, if EA is found to be effective, results from this study can form a solid basis for funding routine establishment of an EA service care model for among symptomatic gallstone diseases patients. Based on the pragmatic nature of the trial, this study will also explore the health economic evaluation of additional acupuncture services against usual care which could facilitate to give an overview for setting up to the integrative medical service.

Aims and Hypotheses to be Tested:

This study aims to evaluate the effectiveness and safety of EA in the treatment of symptomatic gallstone diseases compare with usual care

Hypotheses:

EA could produce greater effects than usual care in treating symptomatic gallstone diseases and increase the rate of excretion.

Objectives

1. To determine whether EA treatment is more effective than usual care in the management of symptomatic gallstone diseases; and
2. To determine whether EA, compared with usual care, can increase clearance rate as confirmed by ultrasonography,
3. To determine the safety of EA in the management of gallstone diseases
4. To explore the health economic assessment of both EA and usual care

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 70 years of age who are diagnosed of gallstone diseases with the last observable ultrasonography.
2. Patients with symptoms such as recurrent biliary colic
3. Wait-listed for elective cholecystectomy or being recommended to have cholecystectomy by surgeons.
4. Largest gallstone size of smaller than 0.8cm.

Exclusion Criteria:

1. Gallstones with the size that cannot be assessed precisely by ultrasound
2. Any gallstone larger than 0.8cm
3. Poor gallbladder ejection fraction computed from Ultrasound-determined fasting and post-prandial gallbladder volumes
4. Contraindication to MRI
5. Patients contraindicated for ERCP
6. Cardiovascular disease with decompensation (New York Heart Association class III or IV)
7. Pregnancy or breastfeeding
8. Alcoholism
9. Intravenous drug users
10. Needle phobia;
11. Unable to respond consistently in trial-out questions of the questionnaire;
12. Refused to provide written informed consent for joining the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of gallstones (excretion of gallstones confirm by ultrasound) | Baseline and 10th week
  Change of ultrasound of baseline and 10th week of gallstones for both treatment group and control group patients.

SECONDARY OUTCOMES:
Change of Gastrointestinal Quality of Life instrument (GIQOLI) | Baseline and 10th week
  The Gastrointestinal Quality of Life Instrument measures the domain based on symptoms related to gastrointestinal tract disorder. GIQLI has four subscales including symptoms, emotions, physical functions, social functions and an item (item 24) related to "troubled by medical treatment". The GIQLI is a 35-item, using a five-point Likert-type scale "from 4 (most desirable option ) to 0 (least desirable option )". The total GIQLI score ranged from 0 to 140, is obtained by adding the score of each answer of the 35 items. Patients with higher scores indicate that patients are with higher QOL. This GIQOLI was validated for gallstone diseases patients. The symptom. GIQOLI will be measured at baseline and 10th week. It measured the quality change of life during the observation period.
132 subjects with Liver function test | Baseline, 5th and 10th week
  132 subjects with Liver function test to measure the liver function across the trial. Blood sample from the liver function includes the blood test for ALT, AST and ALP. Alaine Transaminase (ALT), Asparate Transaminase (AST) and Alkaline Phosphatase (ALP) are important enzyme to reflect the liver function of the body. The monitoring of the liver function tests are very important that may indicate any potential blockage of biliary tree upon during the expel of the gallstone. Therefore the LTF will be assess on baseline, 5th and 10th week.
Clear common bile duct confirm by MRCP | After 10th week if number of gallstones reduced(confirm by ultrasound)
  Number of participants with clearness of ultrasound image. The monitoring of the incidence of common bile duct stone by MRCP to ensure no obstruction of common bile duct in the bilary tree
Number of cases of Serious Adverse Event reported by any subjects | Baseline-10th weeks
  Number of participants with any adverse event including the admission to A&E or reporting of any complications (i.e. acute cholangitis, pancreatitis or etc) will be recorded during the observation period.
Change of EQ-5D | Baseline, 5th week and 10th week
  EuroQol Group - 5 dimensions, EQ-5D, is a utility measure general health on five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The utility can use to measure the quality of life adjusted life years for economic evaluation.This will be measured at baseline, 5th week and 10th week.
  It consists of 5 single-item dimensions including: mobility, self care, usual activities. pain/discomfort, and anxiety/depression. Descriptive data from the 5 dimensions of Part I can be used to generate a health-related quality of life profile for the subject. It measures the quality change of life during the observation period.
Change of EQ VAS | Baseline, 5th week and 10th week
  This is a visual analogue scale, asking to mark health status on the day of the interview on a 20 cm vertical scale with end points of 0 and 100. (0) corresponds to " the worst health you can imagine", and the highest rate (100) corresponds to "the best health you can imagine". Thus the higher marks mean better quality of life, this scale also measures the quality change of life during the observation period.
Change of SF-6D | Baseline, 5th week and 10th week
  Short Form - 6 dimensions, SF-6D is a utility measure general health on two dimensions: physical and mental. The utility can use to measure the quality of life adjusted life years for economic evaluation.The symptoms and Health-related quality of life measured by SF-6D will be measured at baseline, 5th week and 10th week. It measured the quality change of life during the observation period.
  Detail of SF-6D:
  The SF-6D uses 11 questions from the SF-36 to define the six domains (physical functioning, role limitation, social functioning, pain, mental health, and vitality).
  Each domain has between four and six levels. The lower the score the more disability while the higher the score the less disability. Descriptive data from the 6 domains can be used to generate a health-related quality of life profile for the subject, ranging from 0-1, 0 is the worst while 1 is the best.The higher the score, the better the quality of l

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Wong, Dr, Principal Investigator — HKIIM, CUHK
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hksar, China

IPD SHARING:
Plan to Share IPD: Undecided